CLINICAL TRIAL: NCT04959058
Title: EVALUATION OF BRACHIAL PLEXUS IN DIFFERENT ARM POSITIONS BY ELASTOGRAPHY
Brief Title: EVALUATION OF BRACHIAL PLEXUS IN DIFFERENT ARM POSITION
Acronym: ELAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ilker Ince, Associate Professor, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B.30.2.ATA.0.01.00/103
Record Dates: First submitted 2021-05-29; First posted 2021-07-13 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Elasticity Imaging Techniques; Brachial Plexus Injury
Keywords: Brachial plexus, Elastography

STUDY DESIGN:
Intervention Model Description: Measurements will be made in 3 different positions for a participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteer (Other): This study has only one arm for the brachial plexus evaluation with ultrasound
  Interventions: Device: Volunteer

INTERVENTIONS:
Device: Volunteer — An ultrasound machine will be used to calculate the elastographic value of the brachial plexus in three different positions.

SUMMARY:
In daily life,people protect their tissues against ischemia by constantly changing positions. In situations that cause unconsciousness such as anesthesia,people cannot react to the stress or pressure due to immobility.This prolongation of immobility can lead to reversible or irreversible damage to the tissues.Therefore,not careful positioning in patients undergoing surgery can lead to serious complications.Peripheral nerve disorders are common in clinical practice.Electrodiagnostic studies continue to be the gold standard for the evaluation of nerve disorders.Elastography is a technique that measures the elastic properties of tissues as a new ultrasonography technology.Given the histological changes in diseased peripheral nerves, nerve elastography has begun to be studied as a noninvasive way to evaluate changes in nerve tissue composition.Elastography of the peripheral nerves has rarely been studied.

Primary aim in this study is to compare the elastography values of the brachial plexus in different arm and head positions and to contribute to elucidating the mechanism of nerve damage due to position.American Society of Anesthesiologists (ASA) I-II volunteers between the ages of 18-65 will be recruited to the study.The bilateral brachial plexus of each volunteer will be examined.Participants with upper extremity or cervical trauma, muscle weakness,cervical disc herniation or a history of spine or cranial surgery, neuromuscular disease, clinical diagnosis of brachial plexopathies, hyperlipidemia,diabetes mellitus or radiotherapy history in the cervical region,body mass index> 35 will not be taken.Before the procedure, the muscle strength of the upper extremity and cervical muscles will be examined and volunteers with muscle weakness will be excluded from the study.Measurements will be made together by two researchers who have at least 5 years of experience in ultrasonography.Measurements will be made in 3 different positions.When the arm and head are in neutral position, the head is turned to the opposite side and the head is turned to the opposite side, the brachial plexus in the supraclavicular region will be visualized by ultrasonography while the arm is in hyperabduction.The area between the upper boundary and the lower boundary of the plexus will be marked, and the values will be taken 5 times consecutively with the share wave elastography method and the elastic modulus,shear wave velocity will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Volunteers

Exclusion Criteria:

* Upper extremity trauma
* Cervical trauma
* Muscle weakness
* Cervical disc herniation
* History of spine surgery
* Cranial surgery,
* Neuromuscular disease
* Clinical diagnosis of brachial plexopathies
* Hyperlipidemia
* Diabetes mellitus
* Radiotherapy history in the cervical region
* Severely obese volunteers (body mass index> 35 kg / m2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary aim in this study is to compare the baseline measurements of elastography values (kPa-kilopascal) of the brachial plexus in different arm and head positions. | Prestudy will be conducted with volunteers and the measurement will take about 15 minutes per case for three different case position as described in thestudy will be conducted with volunteers and the measurement will take about 15 minutes per subject.

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Ince, Principal Investigator — Ataturk University, Department of Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakaya MA, Darcin K, Ince I, Yenigun Y, Kasali K, Dostbil A. Evaluation of brachial plexus stiffness in different arm and head positions by sonoelastography. Medicine (Baltimore). 2023 Oct 13;102(41):e35559. doi: 10.1097/MD.0000000000035559. PMID 37832128